CLINICAL TRIAL: NCT03832231
Title: Evaluation of Diaphragmatic Function in Mechanically Ventilated Patients With Transient Shear Wave Elastography
Brief Title: Use of Transient Elastogaphy to Assess Diaphragm Function in Mechanically Ventilated Patients
Acronym: Elasto-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180264; 2018-A02311-54 (Other: ANSM)
Record Dates: First submitted 2019-01-11; First posted 2019-02-06 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Ventilator Weaning; Intensive Care Unit
Keywords: Shear wave elastography; Ultrasonography; Transdiaphragmatic pressure; Diaphragmatic function; Mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilator liberating trial (Experimental): The diaphragmatic function of patients undergoing a ventilator liberating trial will be determined with transient shear wave elastography.
  Interventions: Device: Shear Wave Elastography

INTERVENTIONS:
Device: Shear Wave Elastography — Ultrasound technology to assess tissue stiffness

SUMMARY:
Mechanical ventilation is a life-saving treatment that can be associated with diaphragm dysfunction, a potentially deleterious acquired disability. It may be the consequence of disuse - under mechanical ventilation, respiratory muscles are unloaded - or the consequence of muscle overuse because of insufficient unloading. Evaluating diaphragm function is therefore crucial to optimally tailor the ventilator assistance. Measurement of transdiaphragmatic pressure (Pdi) is the reference method to assess diaphragm function but it invasiveness hinders the generalization of its use. Previous studies have reported that ultrasound can quantify diaphragm thickening and that diaphragm thickening fraction (TFdi) is a good marker of diaphragm function. Since diaphragm becomes stiffer when it contracts, the investigators aim at exploring whether the measurement of diaphragm stiffness by transient shear wave elastography would improve the evaluation of diaphragm function with ultrasound.

Therefore, the objectives of the study are to evaluate the performance of transient shear wave elastography applied to the diaphragm to estimate Pdi in mechanically ventilated patients as compared to TFdi and to correlate the changes in elastography derived indices, in TFdi and in Pdi into different ventilatory conditions and during a spontaneous breathing trial. Pdi will be obtained using catheters positioned in patients' stomachs and esophagus and diaphragm stiffness will be assessed by measuring the shear modulus of the diaphragm with a dedicated ultrasound machine (Aixplorer, Ultrasonic). TFdi will be also measured as previously reported. Pdi, TFdi and shear modulus will be measured at the end of each four following 10 minutes-conditions: 1) baseline with initial ventilator settings (set by the physician in charge of patient); 2) 25%-increase in pressure support and initial PEEP; 3) 25%-decrease in pressure support and initial PEEP and 4) initial level of pressure support and ZEEP. Finally, the same measurements will be done at the beginning of a 30 minutes spontaneous breathing trial.

DETAILED DESCRIPTION:
Objective :

The main objective is to correlate ultrasound indices (thickness, thickening, rigidity) to the measurement of transdiaphragmatic pressure in the evaluation of the diaphragmatic function of patients under mechanical ventilation.

Secondary objectives are: 1. Correlate thickening of the diaphragm with Pdi, 2. Correlate diaphragmatic thickening with diaphragmatic stiffness 3. Describe these correlations under different levels of pressure ventilatory support, 4. Describe the evolution of diaphragmatic stiffness, thickening and Pdi pressure during a ventilator liberating trial.

The primary endpoint is the measurement of Pdi. The secondary endpoints are the diaphragm thickening fraction and diaphragm stiffness.

Methods :

The Pdi will be obtained by measuring the esophageal and gastric pressures through nasogastric tube equipped with balloons. The position of each of the balloons will be checked by displaying the esophageal and gastric pressure lines. The intragastric position will be confirmed by mild abdominal compression. The oesophageal position is based on visualization of cardiac artifacts on the pressure pattern and signal deflations related to inspiratory movements. The signals of the esophageal and gastric pressures will be displayed continuously and their resultant - transdiapragmatic pressure - will be automatically calculated in real time by the software. It will also record pressure in the airways at the endotracheal tube.

Patients will be placed in half-sitting position to allow better recognition of the diaphragm. Using the ultrasound system Aixplorer® (Aix en Provence, France V9), equipped with a high resolution probe (6 MHz). The probe will be positioned at the intercostal space above the tenth rib on the right axillary line and directed perpendicular to the diaphragm (apposition zone). The measurements will be performed "offline" and the calculation of the thickening fraction will be performed in blind clinical conditions.

The diaphragmatic elastography will be determined using the same ultrasound system (Aixplorer®, Aix en Provence, France V9, provided with a high resolution probe (SL10-2, central frequency, 6 MHz)). The anatomical approach is the same as the intercostal approach described previously. After finding the diaphragm in B mode, a transition to SWE (elastography) mode will be performed. Three successive measurements will be made on the same region of interest, the average of the three measurements will be retained. The variation of the shear modulus during the inspiratory time will also be calculated post hoc. As for standard ultrasound, records analysis will be performed in blind conditions.

Pdi, ultrasound derived indices and shear wave modulus will be measured under several conditions.

1. At baseline: initial ventilator settings set by the physician in charge of patient
2. 25%-increase in pressure support and initial PEEP during 10 minutes
3. 25%-decrease in pressure support and initial PEEP during 10 minutes
4. initial level of pressure support without PEEP (PEEP = 0) during 10 minutes
5. Measurement of the maximal inspiratory pressure during an inspiratory occlusion maneuver lasting 20 seconds.
6. A 30 minutes Ventilator liberating trial without PEEP nor Pressure Support (CPAP=0)

ELIGIBILITY:
All patients receiving mechanical ventilation and having spontaneous efforts will be eligible if they meet the following criteria:

Inclusion criteria

* Age ≥ 18 years old
* Intubation and mechanical ventilation since 24 hours
* Failure to a first ventilator liberating trial
* nasogastric feeding tube in place
* readiness criteria to undertake a ventilator liberating trial (Boles et al. ERJ 2007)
* patient written consent or next of kin written consent in case of physical inability of the patient to sign the consent form
* french social Health Service registration

Exclusion criteria

* pregnancy
* protective administrative control
* patient's refusal
* contra indications to the insertion of esophageal and gastric balloons
* allergy to topical anesthetic
* impossible weaning (full dependance to mechanical ventilation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Change in transdiaphragmatic pressure | Through patient participation, an average of 1 day
  Reference method to assess diaphragm function computed as the difference between esophageal pressure and gastric pressure

SECONDARY OUTCOMES:
Change in diaphragm thickness and thickening as expressed by the thickening fraction (ratio of the difference between inspiratory and expiratory thickness over expiratory thickness). | Through patient participation, an average of 1 day
  Using the ultrasound system Aixplorer® (Aix en Provence, France V9), equipped with a high resolution probe (6 MHz), anatomical structures will be identify using B-mode. A switch to TM-mode will allow us to measure the thickening fraction. A second switch to shear wave elastography allows to identify an elastography map of the diaphragm and calculate an average of the shear wave modulus.
Change in diaphragm stiffness | Through patient participation, an average of 1 day
  Using the ultrasound system Aixplorer® (Aix en Provence, France V9), equipped with a high resolution probe (6 MHz), anatomical structures will be identify using B-mode. A switch to TM-mode will allow us to measure the thickening fraction. A second switch to shear wave elastography allows to identify an elastography map of the diaphragm and calculate an average of the shear wave modulus.
Success or failure at the spontaneous breathing trial | Through patient participation, an average of 1 day
  Presence of clinical intolerance criteria according to Boles et al. ERJ 20107

CONTACTS AND LOCATIONS:
Overall Officials: Martin DRES, MD, PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France

REFERENCES:
- [Derived] Fosse Q, Poulard T, Nierat MC, Virolle S, Morawiec E, Hogrel JY, Similowski T, Demoule A, Gennisson JL, Bachasson D, Dres M. Ultrasound shear wave elastography for assessing diaphragm function in mechanically ventilated patients: a breath-by-breath analysis. Crit Care. 2020 Nov 27;24(1):669. doi: 10.1186/s13054-020-03338-y. PMID 33246478